CLINICAL TRIAL: NCT02946593
Title: Stroll Safe Outdoor Fall Prevention Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New York University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NewYorkU
Record Dates: First submitted 2016-10-24; First posted 2016-10-27 (Estimated); Last update posted 2022-11-03 (Actual); Status verified 2017-09

CONDITIONS: Accidental Falls

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment (Experimental): Participants in the treatment group will attend a once a week 7-week outdoor fall prevention program that includes didactic presentations, group discussions/problem solving, practice in strategy use, and action planning for safe community mobility.
  Interventions: Behavioral: Stroll Safe outdoor fall prevention program
- Control (Active Comparator): Participants in the control group will receive written information about preventing outdoor falls.
  Interventions: Behavioral: Outdoor fall prevention brochure

INTERVENTIONS:
Behavioral: Stroll Safe outdoor fall prevention program — The structure of the program will model the evidenced-based Lifestyle Re-Design program (Clark et al., 2012). Session 1, 2, 4 & 5 will include a brief didactic presentation about outdoor fall risks and strategy use from the group leader. This will be followed by group discussion/problem solving related to addressing risks. Identified strategies will be recorded on a wipe board and transcribed for group members in order to create handouts. Each 90 minute session will end with action planning, where participants will write down behavioral changes they will implement in the coming week. Session 3 and 6, also 90 minutes, will include outdoor mobility training and practice using strategies discussed in previous sessions. Training sessions will be led by the PI and an assistant. The final session will be a review of risks, strategy use, and reinforcement of behavioral changes in participant's action plans.
  Arms: Treatment
Behavioral: Outdoor fall prevention brochure — The control group participants will be given a written brochure on tips for preventing outdoor falls.
  Arms: Control

SUMMARY:
The purpose of the study is to examine the feasibility of the program and data collection protocol to plan a multisite clinical trial. The program, "Stroll Safe", an outdoor fall prevention program, will take place in the lab space of the New York University occupational therapy department and in the surrounding neighborhood.

Twenty-four people who meet the inclusion criteria will be enrolled after informed consent. Recruitment will include follow up with people who expressed interest in the fall prevention program during a survey study conducted by the PI, and interested members of community-based programs for seniors who have agreed to be community partners for this study. Twelve participants will be assigned to the 7-week program and 12 will receive written information on outdoor fall prevention (control group).

The topics addressed in the once a week, 7-week outdoor falls prevention program, for which a treatment manual has been developed, are based on the results of a survey conducted of community dwelling older adults that identified gaps in knowledge and use of prevention strategies, and the related literature. The program includes pre-set modules, however, participants will be able to voice individual concerns and problem-solve solutions during group discussions. Using an ecological perspective, the Health Belief Model, and problem solving theory as a guide, the intervention will include a didactic component, group problem solving, practical application of strategies, and self-advocacy regarding reporting problems to the city.

Analysis will primarily focus on process measures.Post-intervention, semi-structures interviews will be conducted and analyzed to assess strengths/limitations of the program and participant's attribution of any behavioral changes to the intervention. Although statistical significant is not anticipated in this small feasibility study, repeated measures ANOVA will be used to examine changes in Falls Efficacy Scale-International (FES-I), Outdoor Falls Questionnaire (OFQ) and Falls Behavioral Scale for the Older Person (FaB) scores from pre to post-test for the treatment and control groups. Effect sizes (Cohen's d) will also be calculated. Change in number of stumbles, trips, slips, and falls before and after the program will also be analyzed.

Data will be collected on falls self-efficacy and strategy use at study enrollment (Baseline), after completion of the 7 week program (1st Post-test), and at 2 months post-program completion (2nd Post-test). Participants will be asked to keep daily diaries of stumbles, trips, slips, and falls from the time they enroll in the study until two months following the completion of the program.

ELIGIBILITY:
Inclusion Criteria:

* 55 years of age or older
* English speaking
* Cognitively competent (i.e. a Montreal Cognitive Impairment (MOCA) score >24)
* Able to ambulate outdoors independently with or without an assistive device
* Able to travel independently to the program site
* Have sustained a stumble, trip, slip or fall outdoors within the last year

Exclusion Criteria:

* Younger than age 55
* Living in an institutional setting
* Non-English speaker
* Requiring assistance for outdoor ambulation and/or community mobility
* Cognitively impaired as per MOCA scores
* An active medical, neurological or psychiatric disease that interferes with participation (e.g. stroke, chronic obstructive pulmonary disease requiring supplemental oxygen, Amyotrophic Lateral Sclerosis, and schizophrenia).

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2017-01; Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Change in Outdoor Falls Questionnaire (OFQ) | Baseline, following 7-week program, 2 months post program completion
Change in Falls Behavioral Scale for the Older Person (FaB) | Baseline, following 7-week program, 2 months post program completion
Change in Falls Self-efficacy Scale- International (FES-I) | Baseline, following 7-week program, 2 months post program completion

OTHER OUTCOMES:
Change in Fall diary reports | At baseline, every two weeks until 2 months post program completion

CONTACTS AND LOCATIONS:
Locations (1):
- New York University, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Clark F, Jackson J, Carlson M, Chou CP, Cherry BJ, Jordan-Marsh M, Knight BG, Mandel D, Blanchard J, Granger DA, Wilcox RR, Lai MY, White B, Hay J, Lam C, Marterella A, Azen SP. Effectiveness of a lifestyle intervention in promoting the well-being of independently living older people: results of the Well Elderly 2 Randomised Controlled Trial. J Epidemiol Community Health. 2012 Sep;66(9):782-90. doi: 10.1136/jech.2009.099754. Epub 2011 Jun 2. PMID 21636614
- [Background] Delbaere K, Close JC, Mikolaizak AS, Sachdev PS, Brodaty H, Lord SR. The Falls Efficacy Scale International (FES-I). A comprehensive longitudinal validation study. Age Ageing. 2010 Mar;39(2):210-6. doi: 10.1093/ageing/afp225. Epub 2010 Jan 8. PMID 20061508
- [Background] Chippendale T. Development and validity of the Outdoor Falls Questionnaire. Int J Rehabil Res. 2015 Sep;38(3):263-9. doi: 10.1097/MRR.0000000000000115. PMID 25851838
- [Background] Clemson L, Bundy AC, Cumming RG, Kay L, Luckett T. Validating the Falls Behavioural (FaB) scale for older people: a Rasch analysis. Disabil Rehabil. 2008;30(7):498-06. doi: 10.1080/09638280701355546. PMID 17852314